CLINICAL TRIAL: NCT01377038
Title: Central Pain Mechanisms in Osteoarthritis: A Longitudinal Cohort
Brief Title: OASIS: Osteoarthritis Sensitivity Integration Study
Acronym: OASIS
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Funding
Sponsor: University of Michigan (Other)
Responsible Party: Principal Investigator, Kristine Phillips, Associate Professor, University of Michigan
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2011 HUM00044644
Record Dates: First submitted 2011-06-16; First posted 2011-06-20 (Estimated); Last update posted 2016-10-26 (Estimated); Status verified 2016-10

CONDITIONS: Osteoarthritis; Chronic Pain
Keywords: Osteoarthritis; Chronic pain; Central pain
MeSH Terms: conditions — Osteoarthritis; Chronic Pain

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Duloxetine (Active Comparator): Phenotype assessment prior to and after treatement with duloxetine 20-30 mg oral daily for eight weeks.
  Interventions: Other: Phenotype assessment
- Diclofenac (Active Comparator): Phenotype assessment prior to and after treatment with topical diclofenac four times daily
  Interventions: Other: Phenotype assessment

INTERVENTIONS:
Other: Phenotype assessment — Quantitative sensory testing and patient reported outcome measures used to assess patient pain phenotype

SUMMARY:
The primary objective of this study is to evaluate the relative efficacy of a centrally-acting analgesic (duloxetine) versus a peripherally acting analgesic (topical diclofenac) for pain and associated symptom management in knee osteoarthritis. Secondary objectives include the determination of which self-report and experimental pain measures best differentiate those who respond better to duloxetine than diclofenac.

DETAILED DESCRIPTION:
This is a randomized, blinded, crossover, controlled study design comparing duloxetine and topical diclofenac for osteoarthritis pain.

The study cohort will be individuals who have a confirmed diagnosis of knee osteoarthritis. Subjects will be randomized only after all entry criteria have been met. These individuals will be evaluated at baseline, and then followed longitudinally following enrollment.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with knee osteoarthritis as defined by American College of Rheumatology (ACR) criteria
* Males and females age greater than 50 years at time of screening

Exclusion Criteria:

* History of chronic kidney disease or moderate to severe hepatic impairment
* History of anemia
* Allergy or intolerance of drug intervention
* Inability to participate in outcome measures

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2011-09; Primary Completion 2015-07 (Estimated); Study Completion 2015-07 (Estimated)

PRIMARY OUTCOMES:
Pain | One month

CONTACTS AND LOCATIONS:
Overall Officials: Kristine Phillips, MD, PhD, Principal Investigator — University of Michigan
Locations (1):
- University of Michigan, Ann Arbor, Michigan, United States

REFERENCES:
- [Derived] Murphy SL, Lyden AK, Kratz AL, Fritz H, Williams DA, Clauw DJ, Gammaitoni AR, Phillips K. Characterizing Pain Flares From the Perspective of Individuals With Symptomatic Knee Osteoarthritis. Arthritis Care Res (Hoboken). 2015 Aug;67(8):1103-11. doi: 10.1002/acr.22545. PMID 25580697